CLINICAL TRIAL: NCT05211934
Title: Relationship Between Postoperative Delirium and Heart Function in Valvular Surgery：A Prospective Observational Cohort Study
Brief Title: Relationship Between Postoperative Delirium and Heart Function in Valvular Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Jun Ma, The chief of department of anesthesiology, Beijing Anzhen Hospital
Other Study IDs: 20220101
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Valvular Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The group with delirium
  Interventions: Other: No intervention
- The group without delirium
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Delirium is an acute brain lesion characterized by abnormalities of consciousness, attention, cognition and sensation. Many brain diseases such as stroke, traumatic brain injury and intracranial hypertension can lead to cardiac insufficiency, arrhythmia and heart failure. The incidence of postoperative delirium in patients undergoing cardiac surgery is high. Postoperative delirium is a manifestation of brain function injury. The effect of postoperative delirium on postoperative cardiac function in patients undergoing cardiac surgery is worthy of further discussion.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing valvular surgery
* Age between 60 to 75

Exclusion Criteria:

* Have a history of cerebral infarction before operation
* Cardiac function was seriously impaired before surgery
* Neuropsychiatric disorders were present before surgery

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing valvular surgery in our hospital were selected. The age was 60 years ≤ age ≤75 years, and gender was not limited. According to the occurrence of postoperative delirium, the patients were divided into postoperative delirium group and Non-postoperative delirium group.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
heart function | up to 60 days
  Doses of norepinephrine, epinephrine, dopamine, dobutamine and vasopressin

CONTACTS AND LOCATIONS:
Locations (1):
- Anzhen hospital, Beijing, Beijing, Beijing Municipality, China